CLINICAL TRIAL: NCT04653792
Title: Role Of Pregabalin To Decrease Postoperative Pain In Microdiscectomy: A Randomized Clinical Trial
Brief Title: Role Of Pregabalin To Decrease Postoperative Pain In Microdiscectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ziauddin University (Other)
Responsible Party: Principal Investigator, Shahzaib Riaz Baloch, Senior Resident, Orthopedics Department, Ziauddin University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: preg2020micro
Record Dates: First submitted 2020-11-27; First posted 2020-12-04 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Pain, Nerve; Prolapsed Intervertebral Disc
Keywords: Microdiscectomy; Pregabalin
MeSH Terms: conditions — Neuralgia; Intervertebral Disc Displacement | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Pregabalin (Experimental): Participants received Pregabalin 75mg capsule twice daily from preoperative day to 1 week postoperative
  Interventions: Drug: Pregabalin 75mg
- Pregabalin Placebo (Placebo Comparator): Participants received Pregabalin placebo capsule matching Pregabalin twice daily from preoperative day to 1 week postoperative
  Interventions: Device: Placebo

INTERVENTIONS:
Drug: Pregabalin 75mg — 75 mg capsule
  Other Names: Lyrica (Pregabalin) 75mg
  Arms: Pregabalin
Device: Placebo — 75 mg
  Other Names: Pregabalin placebo
  Arms: Pregabalin Placebo

SUMMARY:
The purpose of this study is to compare the effect of pregabalin in reducing the neuropathic pain in postoperative patients who have undergone single level Microdiscectomy for prolapsed intervetebral lumbar disc.

DETAILED DESCRIPTION:
All patients were informed in detailed regarding the risk and complications and given written and informed consent, coming to our clinics were assessed by one of the senior team members of the spine, patient fulfilling the eligibility criteria were selected and included in the study. One week before the surgery the patients who met the eligibility criteria were randomized in a double-blind manner (participant and investigator) in a ratio of 1:1 into Group-A (Pregabalin 7mg, twice daily) or Group-B (Placebo, twice daily). The pain scores were recorded by VAS and Roland Morris score system on preoperative day compared to the scores on the 1st week postoperative follow-up.

ELIGIBILITY:
Inclusion Criteria:

* All patients with severe CLBP and/or leg pain
* Patients with static or dynamic leg pain
* Patients with leg pain resulting from localized lumbar or lumbosacral segmental instability
* Spinal stenosis at levels L2-S1 or caused by isthmic spondylolisthesis (grade I and II)

Exclusion Criteria:

* Patients with previous lumbar surgery
* Patients allergic to gabapentinoids
* Patients with renal impairments
* Patients who are already on opioids, benzodiazepines, barbiturates, ethanol (alcohol)
* Patient presented with diabetes and other drugs that depress the central nervous system
* Patients who are already on ACE inhibitors as they may enhance the adverse/toxic effect of Pregabalin.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2020-04-17 (Actual); Study Completion 2020-04-17 (Actual)

PRIMARY OUTCOMES:
change from preoperative pain score using a 10 point visual analog scale (VAS pain scale) at 1 week post surgery for PID | Preoperative and one week postoperative
  VAS pain scale is a validated, self-reported instrument assessing average pain intensity over the past 24 hours period. Possible scores being 0 (no pain) and 10 (worst possible pain). Change = (1 week post surgery - preoperative pain)

CONTACTS AND LOCATIONS:
Overall Officials: Shahzaib Riaz, Principal Investigator — Ziauddin University hospital Karachi; Sohail Rafi, FCPS, Study Director — Ziauddin University Hospital Karachi
Locations (1):
- Dr. Ziauddin University Hospital Clifton Campus, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No